CLINICAL TRIAL: NCT03562390
Title: Irinotecan for Advanced and Metastatic Breast Cancer Previously Treated Using Anthracyclines- and Taxanes-containing Regimens: Protocol for a Phase II, Open-label, Single-arm Trial
Brief Title: Irinotecan for Advanced and Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Sun Tao, Principal Investigator, Liaoning Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STao-002
Record Dates: First submitted 2018-06-08; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): 124 women with locally recurrent or metastatic breast cancer who will receive treatment at 17 research centers in Liaoning Province and Heilongjiang Province of China. Irinotecan is administered intravenously on days 1 and 8 of each 3-week cycle.
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Irinotecan — The patients will receive treatment using intravenous irinotecan hydrochloride until the patient develops disease progression or fulfills a withdrawal criterion.

SUMMARY:
This trial aims to evaluate the safety and efficacy of third-line or later irinotecan treatment for locally recurrent or metastatic breast cancer among Chinese patients who have received at least two regimens containing anthracyclines and taxanes.

DETAILED DESCRIPTION:
Anthracyclines and taxanes are the most effective first-line and second-line treatments for breast cancer, although increased usage in early treatment lines can make it difficult to select a third-line or later treatment. This issue is further complicated by the fact that patients with metastatic breast cancer can become resistant to anthracyclines and taxanes. Thus, there are no consistent international guidelines regarding treatment in this setting.

In China, the treatment procedures for metastatic breast cancer follow the National Comprehensive Cancer Network guidelines, which recommend single-drug treatments for recurrent or metastatic disease, which typically involve anthracyclines, taxanes, vinorelbine, gemcitabine, capecitabine, and eribulin. However, there is no standard international recommendation for patients with metastatic breast cancer who have developed resistance to anthracyclines and taxanes, and there are limited options for third-line or later treatment in this setting.

This trial aims to evaluate the safety and efficacy of third-line or later irinotecan treatment for locally recurrent or metastatic breast cancer among Chinese patients who have received at least two regimens containing anthracyclines and taxanes.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-70 years;
* Female patients with histologically or cytologically confirmed breast cancer;
* Patients with locally recurrent or metastatic breast cancer who have been treated with at least two chemotherapy regimens;
* Measurable lesions (based on computed tomography or magnetic resonance imaging) that have a longest diameter of ≥ 10 mm based on the RECIST v1.1 criteria and a shortest lymph node diameter of ≥ 15 mm;
* Eastern Cooperative Oncology Group (ECOG) grade 0-2;
* Life expectancy of ≥ 12 weeks;
* Adequate bone marrow capacity, hepatic functional reserve, and renal functional reserve within 7 days before screening:

Absolute neutrophils count: 1.5 × 109/L Hemoglobin: ≥ 9.0 g/dL;

* Platelet count: ≥ 80 × 109/L Total bilirubin: < 1.5 times the ULN Aspartate and alanine transaminases: ≤ 2.5 times the ULN (≤ 5 times the ULN for liver metastases) Alkaline phosphatase:< 4 times the ULN Serum creatinine: ≤ 1.5 times the ULN
* Women of childbearing age requiring effective contraception;
* Provision of informed consent.

Exclusion Criteria:

* Receiving chemotherapy, radiotherapy, HER2/neu-targeted drugs (including trastuzumab), or hormonal therapy within 3 weeks;
* Breast cancer patients who do not receive local treatment and develop brain and dural metastasis. However, patients will be eligible if corticosteroids for brain and dural metastasis have been withdrawn for at least 4 weeks, if the signs and/or symptoms of brain metastasis have been stable for ≥ 4 weeks, and if imaging findings confirm that the disease is stable between the screening and 4 weeks earlier;
* Severe cardiovascular injury (congestive heart failure of class II or worse based on the New York Heart Association classification), unstable angina, myocardial infarction, or severe arrhythmia during the past 6 months;
* A history of human immunodeficiency virus infection, chronic hepatitis B, or hepatitis C (high viral DNA copyl DNA ti) at the active phase;
* Clinical evidence of other severe active infection;
* Patients with homozygous mutations in UGT1A1*6 and/or UGT1A1*28 (these patients are susceptible to irinotecan-induced diarrhea);
* Patients with allogeneic organ transplants that require immunosuppressive therapy;
* A history of other malignancies within 5 years, except for cured cervical carcinoma in situ or basal cell skin cancer. Women who are pregnant, lactating, or within their childbearing age but not using adequate contraception;
* Drug abuse and medical, psychological, or social conditions that could interfere with the patient's ability to consent or that might affect the study's results;
* Known or suspected being allergy to the studied drug or any other drug administered in the study;
* Any unstable condition that might jeopardize the patient's safety and compliance.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1 year
  The ORR will be calculated based on the number of patients who achieve a complete or partial response divided by the total sample size.

SECONDARY OUTCOMES:
Progression-free survival(PFS) | 1 year
  The PFS interval will be calculated from the start of irinotecan treatment to the first instance of tumor progression, treatment failure, or death from any cause. Overall survival will be calculated from the start of irinotecan treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Sun, Principal Investigator — Cancer Hospital of China Medical University
Locations (1):
- Cancer Hospital of China Medical University, Shenyang, Liaoning, China